CLINICAL TRIAL: NCT02610205
Title: Integrative Care at the Emergency Department
Brief Title: Caring Touch as a Bodily Anchor for Patients After Sustaining a Motor Vehicle Accident
Status: Completed | Type: Observational
Sponsor: Fanny Airosa (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Fanny Airosa, Manager of Nursing Development, Emergency Medicine, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Other Study IDs: Touch-ED
Record Dates: First submitted 2015-11-06; First posted 2015-11-20 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Emergency
Keywords: Caring touch; Tactile massage; Healing touch
MeSH Terms: conditions — Emergencies | interventions — Touch

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Caring touch interventions: The study was conducted as a mixed-methods design. A recruitment of potential study participants was made up from a list of incoming patients arriving at the emergency department following an MVA, and who upon medical examinations were given an injury severity score between 0-3 and subsequently discharged straight home. ISS is a 0-8 point scale rating injury severity, where a rating of 0 indicates no physical injury; 1-3 represents minor physical injuries. The patients were informed about the study by mail during the week after the MVA, and those interested in participating in the caring touch intervention were asked to contact the investigator and subsequently completed a written informed consent form during the first encounter with the therapist.
  Interventions: Other: caring touch

INTERVENTIONS:
Other: caring touch — The caring touch was adjusted to suit each participant and lasted for 20-60 minutes, once a week, for a maximum of eight treatment sessions altogether. The tactile massage, a soft tissue massage, without applying direct pressure or stretching to the muscles. The massage can be described as slow, gentle, structured, circulating movements with the palm of the therapist's hand, during which natural oil, or oil with the fragrance of lavender, was applied. The healing touch was based on an established procedure, during which the therapist applied a light pressure to the feet, ankles, knees, hips, stomach, heart area, arms, throat, forehead and scalp. The participant was fully dressed during the healing touch, as the therapist used her/his hand in different positions on the participant's body.
  Other Names: healing touch; tactile massage

SUMMARY:
The aim of this study was to explore participants´ subjective experiences and perspectives on pain and other factors of importance after an early nursing intervention consisting of "caring touch" (tactile massage and healing touch) for participants subjected to a motor vehicle accident with minor or no physical injuries.

DETAILED DESCRIPTION:
The study was conducted as a longitudinal study, combining qualitative and quantitative perspectives, i.e. a mixed-methods design. The rationale for combining quantitative and qualitative methods was to provide a comprehensive exploration of the research question.Investigators conducted the interviews in a closed meeting room at the hospital, three months after the participant´s first hospital visit. The time span was set to allow the participants to conclude their treatments with caring touch. The interviews, which lasted up to 60 minutes, were conducted in Swedish, digitally recorded and transcribed verbatim by the investigators. An open-ended question was used to initiate the interviews. The quantitative primary outcome was current level of pain measured by VAS, ranging from 0 (no pain) to 100 (worst imaginable pain). Participants rated their current VAS pain at baseline during the initial visit and before and after each treatment session with caring touch, and then again via a postal follow-up after six months. Secondary exploratory outcomes were sense of coherence (SOC), constructed by Antonovsky on the basis of a salutogenic model. The Sense of Coherence scale was of interest since this instrument capture the participants' experiences of comprehensibility, manageability, and meaningfulness which we assumed could be linked to participant recovery. SOC, a 13-item rating scale, developed using the subscales of comprehensibility, manageability, and meaningfulness. Total scores of 21-59 indicate low sense of coherence, 60-74 an average sense of coherence, and 75-91 high sense of coherence. Additionally, the Impact of Event Scale (IES-R) has been well used in previous trauma research and was decided as being an appropriate tool to explore to what extent the participants experienced post-traumatic stress disease. IES-R, 22-item scale shows the degree to which the traumatic experience is felt on a consciousness level, and if the person exhibits avoidant behaviour. The IES-R is based on a 4-point frequency scales (i.e., 0=not at all, 1= a little bit, 2= moderately, 3=quite a bit, and 4=extremely). An average of the total scale sum of 1.8-2.0 indicates post-traumatic stress disorder. The IES-R seems to be a solid measure of post-traumatic phenomena that can augment related assessment approaches in clinical and research contexts. The European Quality of Life (EQ-5D) instrument was employed to explore participants´ health-related quality of life and self-related health. The EQ-5D instrument was selected because of the short-form and that it has been widely used to measure quality of life among the County Councils of Sweden. EQ-5D is a standardized instrument for measuring health outcome. Participants classify their health in terms of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has three levels of severity: (1) no problems, (2) moderate problems, and (3) severe problems. From the sum a number of total 243 combinations of health can be created. Each health combination generates an index value from -0.59 to 1.0, where 1.0 indicates full health. Additionally, the EQ-5D has a visual analogue scale for self-rated health with the anchors at zero (worst imaginable health) up to 100 (best imaginable health).

Data from VAS pain ratings and questionnaires was manually transferred from paper into an electronic database before statistical analysis. Summary characteristics of participants were presented as proportions, mean, median, standard deviation and/or min-max values. Change scores of VAS pain ratings, SOC, IES-R and EQ-5D over time between baseline and follow-up after six months were analysed for patients with complete data. Considering rating scales and ordinal types of data, and the relatively small sample sizes, non-parametric statistical analysis, i.e. the Wilcoxon signed-rank test was employed for assessing change scores over time. All p-value calculations were conducted with a 5% significance level. An additional descriptive analysis was conducted for VAS pain ratings before and after each treatment session with caring touch. Computational software included STATA 13, StataCorp, USA and Microsoft Excel 2011, Microsoft, USA.

ELIGIBILITY:
Inclusion Criteria:

* literate in Swedish and cognitively intact, arriving at the emergency department following an MVA, and who upon medical examinations were given an injury severity score (ISS) between 0-3 and subsequently discharged straight home.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A recruitment of potential study participants was made up from a list of incoming patients, arriving at the emergency department following an MVA, and who upon medical examinations were given an injury severity score (ISS) between 0-3 and subsequently discharged straight home. ISS is a 0-8 point scale rating injury severity, where a rating of 0 indicates no physical injury, 1-3 represents minor physical injuries; and 8 corresponds to a life-threatening injury
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Qualitative interviews | Three months after inclusion
  The interviews, which lasted up to 60 minutes, were conducted in Swedish, digitally recorded and transcribed verbatim by the investigator. An open-ended question was used to initiate the interviews. The interviews were analysed using Systematic Text Condensation (STC), based on Giorgi's psychological phenomenological analysis. The procedure consisted of the following steps: 1) An overview of the data was established, reading through all the interview transcripts; 2) A systematic review of the interviews was made line by line, identifying and sorting meaning units; 3) Meaning units were systematically abstracted and sorted into thematic code groups across individual participants; 4) data was synthesized from the thematic code groups to descriptions and concepts.
Visual analogue scale (VAS) | Change from baseline pain at 6 months
  The quantitative primary outcome was current level of pain measured by VAS, ranging from 0 (no pain) to 100 (worst imaginable pain). Participants rated their current VAS pain at baseline during the initial visit and before and after each treatment session with caring touch, and then again via a postal follow-up after six months. The VAS is a standard instrument for assessing pain that was feasible for the nurses to use in the emergency care setting.

SECONDARY OUTCOMES:
Sense of coherence (SOC) scale | Change from baselines sence of coherence at 6 months
  The Sense of Coherence scale was of interest since this instrument capture the participants' experiences of comprehensibility, manageability, and meaningfulness which we assumed could be linked to participants recovery. SOC, a 13-item rating scale, developed using the subscales of comprehensibility, manageability, and meaningfulness. Total scores of 21-59 indicate low sense of coherence, 60-74 an average sense of coherence, and 75-91 high sense of coherence
Impact of Event Scale (IES-R) | Change from baselines post traumatic stress at 6 months
  The Impact of Event Scale has been well used in previous trauma research and was decided as being an appropriate tool to explore to what extent the participants experienced post-traumatic stress disease. IES-R, 22-item scale shows the degree to which the traumatic experience is felt on a consciousness level, and if the person exhibits avoidant behaviour. The IES-R is based on a 4-point frequency scales (i.e., 0=not at all, 1= a little bit, 2= moderately, 3=quite a bit, and 4=extremely). An average of the total scale sum of 1.8-2.0 indicates post-traumatic stress disorder. The IES-R seems to be a solid measure of post-traumatic phenomena that can augment related assessment approaches in clinical and research contexts.
The European Quality of Life (EQ-5D) | Change from baselines quality of life at 6 months
  The European Quality of Life (EQ-5D) instrument was employed to explore participants´ health-related quality of life and self-related health. The EQ-5D instrument was selected because of the short-form and that it has been widely used to measure quality of life among the County Councils of Sweden. EQ-5D is a standardized instrument for measuring health outcome. Participants classify their health in terms of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has three levels of severity: (1) no problems, (2) moderate problems, and (3) severe problems. From the sum a number of total 243 combinations of health can be created. Each health combination generates an index value from -0.59 to 1.0, where 1.0 indicates full health. Additionally, the EQ-5D has a visual analogue scale for self-rated health with the anchors at zero (worst imaginable health) up to 100 (best imaginable health).

CONTACTS AND LOCATIONS:
Overall Officials: Torkel Falkenberg, PhD, Study Director — Karolinska Institutet

REFERENCES:
- [Derived] Airosa F, Arman M, Sundberg T, Ohlen G, Falkenberg T. Caring touch as a bodily anchor for patients after sustaining a motor vehicle accident with minor or no physical injuries - a mixed methods study. BMC Complement Altern Med. 2016 Mar 22;16:106. doi: 10.1186/s12906-016-1084-2. PMID 27004552